CLINICAL TRIAL: NCT02173860
Title: Strategies for Revascularization in Patients Undergoing Heart Valve Surgery With Concomitant Coronary Artery Disease. AngIography vs Fractional Flow Reserve
Brief Title: Strategies for Revascularization in Patients Undergoing Heart Valve Surgery With Concomitant Coronary Artery Disease
Acronym: SAVE-IT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Portuguese Society of Cardiology (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAVEIT351
Record Dates: First submitted 2014-06-19; First posted 2014-06-25 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Artery Disease; Valvular Heart Disease
Keywords: Coronary artery disease; Valvular heart disease; Fractional flow reserve; Coronary artery bypass surgery; Coronary graft failure or patency
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FFR-guided revascularization (Active Comparator): Patients with valvular heart disease scheduled for elective cardiac surgery and concomitant significant coronary artery disease will have FFR measured with a St. Jude Medical coronary pressure wire across all lesions in vessels pre-specified as suitable for surgical revascularization. If the FFR is ≤0.80, then CABG will be performed. If the FFR is >0.80 then no graft will be placed in that particular vessel. Patients in whom FFR of a particular lesion is not possible can be included if at least one additional lesion is suitable for FFR measurement and grafting.
  Interventions: Procedure: FFR-guided surgical revascularization
- Angio-guided revascularization (Active Comparator): Concomitant CABG will be performed as per clinical routine in all vessels with at least one stenosis > 50%. The vessel should be pre-specified as suitable for surgical revascularization before randomization. An internal mammary graft to the LAD should be attempted in all cases, if possible. Further revascularization strategy is left to the discretion of each center.
  Interventions: Procedure: Angio-guided surgical revascularization

INTERVENTIONS:
Procedure: FFR-guided surgical revascularization
  Other Names: Fractional Flow Reserve-Guided surgical revascularization
  Arms: FFR-guided revascularization
Procedure: Angio-guided surgical revascularization
  Other Names: Coronary artery bypass graft guided by angiographic-only assessment of severity stenosis
  Arms: Angio-guided revascularization

SUMMARY:
The purpose of this study is to determine whether, in patients undergoing elective valvular heart surgery, revascularization of concomitant coronary artery disease (CAD) guided by FFR (Fractional flow reserve) would be superior to standard angiography-guided-revascularization approach on major efficacy and safety outcomes

DETAILED DESCRIPTION:
The SAVE-IT trial is a multicenter, international, randomized, controlled, superiority trial. Patients scheduled to undergo elective valvular heart surgery will be screened for presence of concomitant coronary artery disease (CAD) by invasive coronary angiography. Patients with a stenosis > 50% in at least one epicardial vessel (excluding left main) considered suitable for surgical revascularization will be randomized to FFR guided- or standard angiography-guided surgical revascularization. A proportion of patients with no concomitant CAD will be followed in a parallel registry

Baseline clinical, laboratory, electrocardiographic and echocardiographic data will be obtained. Coronary anatomy severity will be assessed by quantitative coronary angiography (QCA) and Synergy between Percutaneous Coronary Intervention with Taxus and Cardiac Surgery (Syntax) score. Surgical risk will be assessed by Euroscore. Patients randomized to FFR-guided arm will have functional severity of the angiographic stenosis assessed by a St. Jude Medical coronary pressure wire measurement under hyperemic conditions using intravenous or intracoronary adenosine administration. If the FFR is ≤0.8 then a graft will be placed distal to the coronary stenosis. If the FFR is >0.8 no grafting will be performed to the epicardial vessel containing the stenosis. Patients will receive cardiac surgery no later than 8 weeks after randomization.

Peri-operative data will be collected. Clinical follow-up data will be collected at 1, 6 and 12 month after surgery. Graft patency at 12 months will be assessed by cardiac computed angiography (CCTA) for all patients who received at least one graft, except if an invasive coronary angiography has been performed in the preceding 3 months based on clinical grounds.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Severe heart valve disease with indication for an elective cardiac with a St. Jude Medical Heart Valve
* Concomitant significant CAD (at least one epicardial vessel with a stenosis> 50%)
* Willing and able to provide informed written consent

Exclusion Criteria:

* Previous CABG
* Angiographic significant lesion involving left main lesion (patient is still eligible if right coronary artery is candidate for FFR measurement and surgical revascularization)
* All lesions in extremely tortuous or calcified coronary vessels
* Recent myocardial infarction (< 30 days)
* Cardiogenic shock or clinical instability (i.e. NYHA 4, uncontrolled arrhythmias, unexplained hypotension severe bradycardia or any other medical condition considered as a sign of instability by the assisting physician)
* Severe left ventricular dysfunction (EF < 35%)
* Pregnant or are planning to become pregnant during the duration of the investigation
* Chronic renal dysfunction as defined as estimated glomerular filtration rate < 60 ml/min
* Life expectancy < 12 months
* Currently participating in any other clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2016-07; Primary Completion 2021-01 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
MACCE | 12 months
  Composite endpoint of death, nonfatal myocardial infarction, unplanned revascularization and stroke at 12 months. Subjects who die or are lost to follow up before 1 year will be censored at their last recorded activity.
Graft failure | 12 months
  Graft patency as assessed by CCTA scheduled at 12 months. Graft status can also be assessed by invasive coronary angiography if clinically indicated.

SECONDARY OUTCOMES:
MACCE | 1 month
  death, nonfatal myocardial infarction, unplanned revascularization and stroke
MACCE | 6 months
  death, nonfatal myocardial infarction, unplanned revascularization and stroke

OTHER OUTCOMES:
Post operative atrial fibrillation rate | Participants will be followed for the duration of hospital stay, an expected maximum of 4 weeks
  Occurrence of any documented episode of symptomatic or asymptomatic episode of atrial fibrillation
Post operative ICU stay | participants will be followed for the duration of hospital stay, an expected maximum of 4 weeks
  From cardiac surgery end to transfer to intermediate care unit or ward. Measured in hours.
Hospitalization period | expected average of ten days
  From cardiac surgery to hospital discharge. Measured in days.From date of cardiac surgery until the date of first hospital discharge assessed up to 8 weeks
Total circulatory bypass time | expected maximum of 300 minutes
  measured in minutes
Total cross-clamp time | expected maximum of 300 minutes
  measured in minutes
Acute renal injury | to post-operative day 4
  Percentage decline in glomerular filtration rate at post-operative day 4 as compared to pre-operative glomerular filtration rate
Blood transfusion | participants will be followed for the duration of hospital stay, an expected maximum of 4 weeks
  Number of units of red blood cells transfused.
Duration of mechanical ventilation | participants will be followed for the duration of hospital stay, an expected maximum of 4 weeks
  Total duration of mechanical ventilatory support. Repeated intubation will be included
Time to inotropic weaning | participants will be followed for the duration of hospital stay, an expected maximum of 4 weeks
  Total time spent with inotropic support. Recurrent use will be quantified
Use of intra-aortic balloon pump (IABP) | participants will be followed for the duration of hospital stay, an expected maximum of 4 weeks
  Number of patients requiring mechanical hemodynamic support with IABP
Anginal status | 12 months
  Symptomatic status as defined canadian cardiac society (CCS) anginal status score
Heart failure symptoms | 12 months
  Symptomatic status as defined per New York Heart Association (NYHA) score

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Ramos, MD, Principal Investigator — Hospital Santa Marta, Centro Hospitalar Lisboa Central; Sergio Batista, MD, Principal Investigator — Hospital Fernando da Fonseca; Luis Raposo, MD, Principal Investigator — Hospital de Santa Cruz, Centro Hospitalar de Lisboa Central; Emanuele Barbato, PhD, Principal Investigator — Olzv-Aalst Clinic; Colin Berry, PhD, Principal Investigator — Golden Jubilee National Hospital
Locations (1):
- Hospital Santa Marta, centro Hospitalar Lisboa Central, Lisbon, Lisbon District, Portugal